CLINICAL TRIAL: NCT01283659
Title: Computed Tomographic Coronary Angiography for Heart Failure Patients (CTA -HF) Project I-C of Imaging Modalities to Assist With Guiding Therapy and the Evaluation of Patients With Heart Failure (IMAGE-HF)
Brief Title: IMAGE-HF Project I-C: Computed Tomographic Coronary Angiography for Heart Failure Patients
Acronym: CTA-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); The Finnish Funding Agency for Technology and Innovation (TEKES) (Other Government)
Responsible Party: Principal Investigator, Rob Beanlands, Rob S. Beanlands, MD, FRCPC, Chief of Cardiology, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Project I-C; CIF-99470 (Other Grant/Funding Number: Canadian Institutes of Health Research); NCT01622985 (obsolete NCT alias)
Record Dates: First submitted 2011-01-20; First posted 2011-01-26 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure
Keywords: computed tomographic angiography; coronary angiogram; cost effectiveness; QoL; Heart failure; diagnostic accuracy; prospective comparative effectiveness randomized clinical trial
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard imaging (coronary angiography) (Active Comparator): Subjects will undergo a coronary angiogram as planned by their attending doctor
  Interventions: Other: Standard Imaging
- Advanced imaging (CTA) (Active Comparator): Subjects will undergo a CTA scan first. Based on the CTA results, subjects may or may not proceed to coronary angiography. CTA results will be reviewed by the attending physician.
  Interventions: Other: Advanced Imaging

INTERVENTIONS:
Other: Standard Imaging
  Other Names: Coronary Angiography
  Arms: Standard imaging (coronary angiography)
Other: Advanced Imaging
  Other Names: Coronary Computed Tomographic Angiography
  Arms: Advanced imaging (CTA)

SUMMARY:
Background: The prevalence of heart failure (HF) is rapidly rising in industrialized and developing countries. Though invasive coronary angiography (ICA) remains the gold standard for anatomical assessment of coronary arteries and luminal stenoses in these patients, alternatives have been sought. Computed tomographic coronary angiography (CTA) has emerged as an accurate non-invasive diagnostic tool for CAD and has been demonstrated to have prognostic value. Whether or not CTA can be used in patients with HF for diagnosis and to guide patient investigations and management is unknown. Acknowledging the aging population in industrialized counties, the increasing burden of healthcare and growing prevalence of HF, there is a need to identify non-invasive diagnostic tests that are cost-effective, readily available, safe and of sufficient accuracy to risk stratify patients and guide investigations and management.

Methods: The proposed randomized controlled trial (RCT) will evaluate the clinical utility of computed tomographic coronary angiography (CTA) and investigate its potential benefit on resource utilization and health economics in patients with progressive or newly diagnosed heart failure (HF) of unknown etiology (i.e. ischemic versus non- ischemic) or in whom the definition of coronary anatomy is required for diagnosis and management. The experimental algorithm will be compared to invasive coronary angiography (ICA)

Analysis of composite clinical events and major adverse cardiac events will be performed to determine the impact of these strategies upon patient outcomes. Accuracy of CTA in detection of coronary anatomy and obstruction will be assessed in patients undergoing ICA. It is expected that CTA will be a more cost-effective strategy for diagnosis; yielding similar outcomes with fewer procedural risks and improved resource utilization.

DETAILED DESCRIPTION:
Hypotheses Primary Hypothesis: Compared to ICA, a diagnostic strategy algorithm using CTA for patients with HF of unknown etiology or where the definition of coronary anatomy is required for diagnosis and management, will result in a reduction in downstream resource utilization and per patient cost.

Secondary Hypotheses: I) Compared to standard care, a strategy that uses CTA will achieve: a) similar composite clinical events (CCE), quality of life (QoL), major adverse cardiac events (MACE); b) a lower rate of procedure related complications (death, MI, stroke, vascular complications, severe allergic reactions; contrast nephropathy); c) a lower rate of normal ICA. II) Using patient-based analysis and vessel-based analysis, CTA has very good agreement with ICA among patients with HF in the CTA arm who proceed to ICA.

Objectives The primary objective is to understand the role of CTA in patients with HF of unknown etiology. We propose a prospective randomized study of 250 patients to examine the potential impact of CTA compared to ICAon resource utilization and health care costs in patients with HF with unknown CAD status.

Secondary objectives are to: compare CCE, QoL and MACE in the CTA and ICA arms. Radiation exposure and safety in both groups will also be assessed.

Trial design The proposed trial is a multicentre randomized controlled trial of 250 patients. In addition, a retrospective review of the current CTA and ICA databases at the University of Ottawa Heart Institute will be conducted to identify an additional cohort of patients (200-400) where the imaging modality decision has already been made. These patients are not eligible for randomization, but will be entered into a registry.

Trial interventions - Randomization All HF patients requiring investigation to determine the etiology of HF (ischemic versus non-ischemic) will be screened for the study. Patients will be randomized to the investigation arm CTA or ICA. Patients will be stratified according to recruitment site and pre-test probability for obstructive CAD. A stratified block (varying sizes) randomization scheme will be used. Within each strata, patients will be randomized with varying block sizes into the two study groups. A central randomization scheme (envelope), which will ensure concealment, will be used and the local research co-ordinator will perform patient assignments. The randomization scheme will be generated by a statistician using a SAS macro.

ELIGIBILITY:
Inclusion Criteria Eligible HF patients with an admission to hospital or emergency room for heart failure

OR

a documented history of left ventricular dysfunction (LVEF <50%)

OR

a documented history of Class ll-lV heart failure symptoms, in the preceding 12 months prior to enrollment, in whom the diagnosis of CAD is uncertain or the definition of coronary anatomy is required for diagnosis and management.

Exclusion criteria:

1. Age < 18 years or lack of consent,
2. Renal Insufficiency (GFR < 45 ml/min);
3. Allergy to intravenous contrast agents;
4. Contraindication to radiation exposure (e.g. pregnancy);
5. Uncontrolled HR at time of scan (as per local clinical routine)
6. History of revascularization (CABG or PCI);
7. Atrial fibrillation, frequent atrial or ventricular ectopy (> 1 / minute);
8. Unable to perform 20 second breath-hold;
9. CTA or ICA within the preceding 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2011-02; Primary Completion 2017-12 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Resource Utilization | 3 and 12 months
  Primary Outcome Measure: Resource Utilization: will be measured as detailed in Appendix A. Cost: the incremental cost of the diagnostic strategy using CTA will be the primary endpoint and will be estimated through regression methods.

SECONDARY OUTCOMES:
Clinical Endpoints | 3 and 12 months
  CCE, LV Function, QoL, and Safety: will measured.
CTA Accuracy | Baseline
  CTA Accuracy: To address one of the secondary hypotheses: the accuracy in the cohort of patients with CTA undergoing ICA (~ n=100) diagnostic test characteristics (sensitivity, specificity, predictive values and likelihood ratios) will be determined and reported with 95% confidence intervals (CI).

CONTACTS AND LOCATIONS:
Overall Officials: Rob SB Beanlands, MD, FRCP C, Study Director — University of OttawaHeart Institute; Benjamin Chow, MD, FRCP C, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (15):
- Canada (12):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Manitoba, Winnipeg, Manitoba
  - Dalhousie University, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - University of Laval, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec
- Finland (3):
  - Helsinki University Central Hospital,, Helsinki
  - University of Kuopio, Kuopio
  - University of Turku, Turku

REFERENCES:
- [Background] Paterson DI, OMeara E, Chow BJ, Ukkonen H, Beanlands RS. Recent advances in cardiac imaging for patients with heart failure. Curr Opin Cardiol. 2011 Mar;26(2):132-43. doi: 10.1097/HCO.0b013e32834380e7. PMID 21297464
- [Background] Chow BJ, Green RE, Coyle D, Laine M, Hanninen H, Leskinen H, Rajda M, Larose E, Hartikainen J, Hedman M, Mielniczuk L, O'Meara E, deKemp RA, Klein R, Paterson I, White JA, Yla-Herttuala S, Leber A, Tandon V, Lee T, Al-Hesayen A, Hessian R, Dowsley T, Kass M, Kelly C, Garrard L, Tardif JC, Knuuti J, Beanlands RS, Wells GA; IMAGE-HF Investigators. Computed tomographic coronary angiography for patients with heart failure (CTA-HF): a randomized controlled trial (IMAGE HF Project 1-C). Trials. 2013 Dec 26;14:443. doi: 10.1186/1745-6215-14-443. PMID 24369097
- [Derived] Chow BJW, Coyle D, Hossain A, Laine M, Hanninen H, Ukkonen H, Rajda M, Larose E, Hartikainen J, Mielniczuk L, Kass M, Connelly KA, O'Meara E, Garrard L, Bishop H, Small G, Hedman M, Coyle K, Yla-Herttuala S, Knuuti J, Wells GA, Beanlands RS; IMAGE-HF Investigators. Computed tomography coronary angiography for patients with heart failure (CTA-HF): a randomized controlled trial (IMAGE-HF 1C). Eur Heart J Cardiovasc Imaging. 2021 Aug 14;22(9):1083-1090. doi: 10.1093/ehjci/jeaa109. PMID 32588042